CLINICAL TRIAL: NCT07260032
Title: Using Advanced Imaging to Determine the Benefits of Exercise on Cardiovascular Risk in PTSD
Brief Title: Determining the Benefits of Exercise on Cardiovascular Risk in PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Antonia V. Seligowski, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P003032
Record Dates: First submitted 2024-12-04; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: PTSD; Cardiovascular Disease; Cardiovascular Disease Risk Factors
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Other)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The exercise program will consist of specifically designed activities to place a gradually increasing workload on the cardiovascular system.

SUMMARY:
The purpose of this study is to use a non-invasive imaging technique called positron emission tomography/magnetic resonance imaging (PET/MRI) to investigate the effects of exercise on brain activity and arterial (blood vessel) inflammation in people with PTSD symptoms and evidence of or elevated risk for artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Trauma exposure
* PTSD symptoms
* Subclinical atherosclerotic CVD (e.g., coronary, cerebrovascular, or peripheral arterial plaque or calcifications on imaging), clinical atherosclerotic CVD (e.g., myocardial infarction or revascularization), or increased risk for atherosclerotic CVD (i.e., >2 of hypertension, diabetes mellitus, hyperlipidemia, and active smoking)
* Ability to understand and sign informed consent

Exclusion Criteria:

* History of stroke, brain surgery, or seizure
* Use of certain CVD medications (e.g., beta-blockers, high-intensity statins [e.g., rosuvastatin 20/40 mg and atorvastatin 40/80 mg], PCSK-9 inhibitors)
* Psychiatric or cardiovascular medication change within 4 weeks (i.e., stable regimen is allowed)
* Unstable blood pressure or cardiac arrhythmia
* Currently in a supervised or graduated exercise program
* Neurological or systemic inflammatory disease/current systemic anti-inflammatory therapy
* Moderate/severe alcohol/substance use disorder
* Current mania/psychosis
* Weight >300 lbs.
* Claustrophobia
* Pregnancy
* Metal implants
* Uncontrolled hyperglycemia (HgbA1c>7.5%)
* Subjects who have had significant radiation exposure as part of research (>2 nuclear tests, computed tomography images, or fluoroscopic procedures) during the preceding 12-months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Pre-treatment; Post-treatment (12-16 weeks after pre-treatment visit)
  10-minute resting heart rate will be measured in beats per minute and collected from electrocardiogram (ECG)
Blood pressure | Pre-treatment; Post-treatment (12-16 weeks after pre-treatment visit)
  Systolic and diastolic blood pressure
Heart rate variability | Pre-treatment; Post-treatment (12-16 weeks after pre-treatment visit)
  10-minute resting heart rate variability will be measured using heart rate R-peak interval times collected from electrocardiogram (ECG)
Arterial inflammation | Pre-treatment; Post-treatment (12-16 weeks after pre-treatment visit)
  Aortic and carotid arterial inflammation will be based on uptake of 18F-fluorodeoxyglucose during positron emission tomography in these sites
Bone marrow inflammation | Pre-treatment; Post-treatment (12-16 weeks after pre-treatment visit)
  Bone marrow inflammation will be based on uptake of 18F-fluorodeoxyglucose during positron emission tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No